CLINICAL TRIAL: NCT00365092
Title: Early Otitis and Literacy and Attention at 9 to 11 Years
Brief Title: Middle Ear Disease Before Age 3, Treatment With Ear Tubes, and Literacy and Attentional Abilities at Ages 9 to 11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD042080 (NIH)
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2006-08

CONDITIONS: Otitis Media; Middle Ear Effusion
Keywords: Insertion of tympanostomy tubes; Otitis media with effusion; Child development; Literacy; Attention; Middle-ear effusion; Educational status; Behavior; Social behavior; Achievement
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion; Literacy; Behavior; Social Behavior

INTERVENTIONS:
Procedure: Insertion of tympanostomy tubes

SUMMARY:
Middle-ear disease (infection and fluid) is the most common illness in young children after the common cold. Because hearing loss accompanies middle-ear disease, and because early life is a period of rapid development, concern has existed that sustained periods of middle-ear disease might cause lasting impairments of learning, speech development, language development, or behavior and social adjustment. Earlier phases of this research found that the insertion of ear tubes in children younger than 3 years of age with persistent middle-ear disease did not affect their development at 3, 4, or 6 years of age. This study examines the children's literacy, attention, and related abilities at 9 to 11 years of age.

DETAILED DESCRIPTION:
Concern has long existed that persistent otitis media in young children, because of the associated conductive hearing loss, can result in lasting impairments of the children's development. Accordingly, myringotomy with insertion of tympanostomy tubes has often been undertaken in such children in order to promptly restore hearing to normal. However, evidence concerning developmental effects of persistent early-life otitis media has been inconclusive, and evidence that tube insertion in affected children influences their development favorably has been lacking. From a previous study we reported that among a cohort of children younger than three years of age with persistent effusion, prompt as compared with delayed insertion of tympanostomy tubes did not result in improved developmental outcomes in the children at three, four, and six years of age. The purpose of the present study was to assess developmental outcomes in the same children at nine to eleven years of age.

Beginning in 1991, we enrolled 6350 healthy infants less than 62 days of age and evaluated them at least monthly until they reached three years of age. We randomly assigned 429 of the children who developed persistent middle-ear effusion before reaching that age to have tympanostomy tubes inserted either promptly or up to nine months later if effusion persisted. At three, four, and six years of age we systematically assessed the children's cognitive, language, speech, and psychosocial development. In the present study, using a standardized battery of assessments, we evaluated literacy, attentional abilities, social skills, and academic achievement in 391 of these children at nine to eleven years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, less than 62 days of age at enrollment

Exclusion Criteria:

* birth weight less than 5 lb (2268 g)
* small for gestational age
* history of neonatal asphyxia or other serious illness
* major congenital abnormality or chronic illness
* multiple birth
* sibling enrolled in the study
* in foster care or adopted before enrollment
* mother dead, seriously ill, a known drug or alcohol abuser before enrollment
* mother judged by study personnel to be too limited socially or intellectually to give informed consent or adhere to the study protocol
* mother less than 18 years of age
* English not the only household language

Ages: 0 Years to 61 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400
Dates: Start 2002-04; Study Completion 2005-03

PRIMARY OUTCOMES:
All measures at 9 to 11 years of age:
Woodcock Reading Mastery Tests-Revised-Normative Update
Number of words in a grade-level passage read correctly in one minute
Dictation Samples subtest of the Woodcock-Johnson III Tests of Achievement, Standard Battery
Writing Samples subtests of the Woodcock-Johnson III Tests of Achievement, Standard Battery
Elision and Rapid Letter Naming subtests of the Comprehensive Test of Phonological Processing
Children's version of the Hearing in Noise Test
Disruptive Behavior Disorders Rating Scale
Child Behavior Checklist, parent report
Child Behavior Checklist, teacher report
Impairment Rating Scales, parent report
Impairment Rating Scales, teacher report
Computerized visual continuous performance test
Computerized auditory continuous performance test
Wechsler Abbreviated Scale of Intelligence
Computational subtest of the Woodcock-Johnson III Tests of Achievement, Standard Battery

CONTACTS AND LOCATIONS:
Overall Officials: Jack L Paradise, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Paradise JL, Campbell TF, Dollaghan CA, Feldman HM, Bernard BS, Colborn DK, Rockette HE, Janosky JE, Pitcairn DL, Kurs-Lasky M, Sabo DL, Smith CG. Developmental outcomes after early or delayed insertion of tympanostomy tubes. N Engl J Med. 2005 Aug 11;353(6):576-86. doi: 10.1056/NEJMoa050406. PMID 16093466
- [Background] Paradise JL, Dollaghan CA, Campbell TF, Feldman HM, Bernard BS, Colborn DK, Rockette HE, Janosky JE, Pitcairn DL, Kurs-Lasky M, Sabo DL, Smith CG. Otitis media and tympanostomy tube insertion during the first three years of life: developmental outcomes at the age of four years. Pediatrics. 2003 Aug;112(2):265-77. doi: 10.1542/peds.112.2.265. PMID 12897272
- [Background] Paradise JL, Feldman HM, Campbell TF, Dollaghan CA, Colborn DK, Bernard BS, Rockette HE, Janosky JE, Pitcairn DL, Sabo DL, Kurs-Lasky M, Smith CG. Early versus delayed insertion of tympanostomy tubes for persistent otitis media: developmental outcomes at the age of three years in relation to prerandomization illness patterns and hearing levels. Pediatr Infect Dis J. 2003 Apr;22(4):309-14. doi: 10.1097/01.inf.0000059764.77704.55. PMID 12690269
- [Background] Paradise JL, Feldman HM, Campbell TF, Dollaghan CA, Colborn DK, Bernard BS, Rockette HE, Janosky JE, Pitcairn DL, Sabo DL, Kurs-Lasky M, Smith CG. Effect of early or delayed insertion of tympanostomy tubes for persistent otitis media on developmental outcomes at the age of three years. N Engl J Med. 2001 Apr 19;344(16):1179-87. doi: 10.1056/NEJM200104193441601. PMID 11309632
- [Derived] MacKeith S, Mulvaney CA, Galbraith K, Webster KE, Connolly R, Paing A, Marom T, Daniel M, Venekamp RP, Rovers MM, Schilder AG. Ventilation tubes (grommets) for otitis media with effusion (OME) in children. Cochrane Database Syst Rev. 2023 Nov 15;11(11):CD015215. doi: 10.1002/14651858.CD015215.pub2. PMID 37965944
- [Derived] Paradise JL, Feldman HM, Campbell TF, Dollaghan CA, Rockette HE, Pitcairn DL, Smith CG, Colborn DK, Bernard BS, Kurs-Lasky M, Janosky JE, Sabo DL, O'Connor RE, Pelham WE Jr. Tympanostomy tubes and developmental outcomes at 9 to 11 years of age. N Engl J Med. 2007 Jan 18;356(3):248-61. doi: 10.1056/NEJMoa062980. PMID 17229952